CLINICAL TRIAL: NCT01378871
Title: Phase II Study of Therapy With IMTOX-25 in Adults With Refractory/Relapsed Cd25 Positive Adult T Cell Leukemia/Lymphoma
Brief Title: A Phase II Study Of Imtox-25 In Adults With Refractory/Relapsed Cd25 Positive Adult T Cell Leukemia/Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: IND withdrawn
Sponsor: Amit Verma (Other)
Responsible Party: Sponsor-Investigator, Amit Verma, Professor, Oncology, Albert Einstein College of Medicine
Organization: Albert Einstein College of Medicine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-530
Record Dates: First submitted 2011-05-12; First posted 2011-06-23 (Estimated); Results first posted 2023-06-09 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-05

CONDITIONS: Adult T Cell Leukemia; Adult T Cell Lymphoma
Keywords: T Cell; T-Cell; Leukemia; Lymphoma; Leukemia/Lymphoma; ATL
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia; Lymphoma | interventions — RFT5-SMPT-dgA immunotoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Antibody Therapy (Experimental): Treatment with Imtox-25 intravenously over 4 hours every other day for 4 doses. Hospital admission is required during this treatment.
  Interventions: Drug: IMTOX-25

INTERVENTIONS:
Drug: IMTOX-25 — This agent is supplied as a sterile solution at 0.5 mg/ml. Thus a vial with 5 mL contains 2.5 mg IMTOX-25
  IMTOX-25 is an immunotoxin. It is an antibody that is bound to a piece of the poison ricin. This antibody have been shown to bind to leukemia cells and kill them because of the ricin.
  15 mg/m²/cycle IV. The calculated total dose for the cycle will be divided by four and given on Days 1, 3, 5 and 7.
  Other Names: RFT5-dgA

SUMMARY:
This clinical trial will be a multicenter phase II fixed-dose trial in which a minimum of 10 patients with immunophenotypically confirmed ATL with at least 50% of the blasts expressing CD25 as measured by flow cytometry at relapse, will receive Imtox-25. Patients are eligible for repeat courses of treatment every two weeks if they do not experience a dose limiting toxicity (DLT) as defined in Section 5.2 and do not have a HAMA/HARA level > 1 μg/ml. The treatment will be administered in the in-patient setting. If no response is observed among the initial 9 patients, the study would be terminated early and declared negative; if at least one response is observed, accrual would continue to a total of 17 evaluable patients (total study size=19 to account for 10% of the patients being unevaluable for any reason).

DETAILED DESCRIPTION:
Adult T Cell Leukemia/Lymphoma (ATL) is a lymphoproliferative disease associated with HTLV-1 infection, characterized by circulating malignant cells expressing the IL-2 receptor (CD25). Prognosis for patients with ATL remains poor despite advances in chemotherapy, with survival in leukemic patients ranging from six months to less than one year. Novel agents that are potent and specific for the tumor cells are urgently needed to improve overall survival and decrease toxicity in this dismal disease. One therapeutic approach would be to use immunotoxins (ITs). ITs utilize a potent toxin linked to a targeting moiety designed to maximize drug delivery to the tumor cells, thus avoiding the nonspecific toxicity of conventional chemotherapeutic agents. Imtox-25 is constructed using the RFT5 murine monoclonal antibody (Mab) coupled to deglycosylated ricin-A chain (dgA) via the heterobifunctional, thiol-containing crosslinker, 4[(succinimidyloxy) carbonyl]-ƒÑ-methyl-ƒÑ-(2 pyridyldithio) toluene (SMPT). Phase I and II clinical studies with Imtox-25 (RFT5.dGA) have been shown safety and efficacy in adult patients with Hodgkin¡¦s disease and a recommended Phase II dose has been established.. In vitro experiments using ATL cell lines and in vivo studies in a murine xenograft model have demonstrated significant activity of Imtox-25 in this disease. Based on these results, the investigators propose to conduct a phase II trial utilizing Imtox-25 in adults with relapsed or refractory ATL.

ELIGIBILITY:
Inclusion Criteria:

* Age > 17 years inclusive at the time of original diagnosis of HTLV-1 associated ATL.
* Histologic verification of ATL and HTLV-1 sero-positivity at diagnosis and either evidence of relapse/refractory disease based on a Bone Marrow/Peripheral Blood examination or evidence by flow cytometry.
* Disease refractory to conventional CHOP based therapy or transplantation or deemed ineligible for salvage by transplantation.
* Presence of CD25 on at least 50% of the lymphoblasts obtained via BMA or peripheral blood as determined by flow cytometry.
* ECOG performance status 2.
* Life expectancy of > 2 months.
* Patients must have recovered from effects of prior therapy. At least 2 weeks should have elapsed since the last dose of chemotherapy (4 weeks in the case of nitrosourea-containing therapy). Steroids are considered as chemotherapy. However, if the patient has recovered from the side effects of prior therapy and has had a > 50% rise in peripheral blast count, they are immediately eligible. The 50% rise in peripheral blast count must be calculated as follows. The sample for the baseline peripheral blast count must have been taken at least 24 hours after the end of chemotherapy. The sample for the peripheral blast count that is increased by 50% of the baseline peripheral blast count may be taken at any subsequent time. A second peripheral blast count confirming the 50% rise is recommended.
* No hematopoietic limitations as patients with relapsed leukemia routinely have pancytopenia and ITs have not demonstrated hematopoietic toxicity.
* Adequate renal function defined as a serum creatinine 1.5 x normal range.
* Adequate liver function defined as a total bilirubin 1.5 x normal range and SGOT (AST) or SGPT (ALT) 1.5 x normal range.
* Adequate cardiac function defined as a shortening fraction of 27% by echocardiogram, or ejection fraction of 35-40% by MUGA scan.
* Adequate pulmonary function defined as no evidence of dyspnea at rest.
* Normal neurological exam.
* Patient and/or legal guardian must sign a written informed consent.
* All institutional, FDA, and NCI requirements for human studies must be met.

Exclusion Criteria:

* Presence of leukemic or infectious pulmonary parenchymal disease or presence of a pulmonary effusion by chest x-ray.
* Presence of CNS involvement with leukemia.
* History of documented seizure disorder or abnormal neurological examination.
* Human anti-mouse (HAMA) levels of < 1 μg/ml.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2010-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samir Parekh, MD, Principal Investigator — Montefiore Medical Center
Locations (6):
- United States (6):
  - Albert Einstein Cancer Center at Albert Einstein College of Medicine, The Bronx, New York
  - Albert Einstein Cancer Center, The Bronx, New York
  - Albert Einstein Comprehensive Cancer Center, The Bronx, New York
  - Montefiore Medical Center, The Bronx, New York
  - Albert Einstein Clinical Cancer Center, The Bronx, New York
  - Montefiore Medical Center-, The Bronx, New York

REFERENCES:
- [Background] Taylor GP, Matsuoka M. Natural history of adult T-cell leukemia/lymphoma and approaches to therapy. Oncogene. 2005 Sep 5;24(39):6047-57. doi: 10.1038/sj.onc.1208979. PMID 16155611
- [Background] Waldmann TA, Goldman CK, Bongiovanni KF, Sharrow SO, Davey MP, Cease KB, Greenberg SJ, Longo DL. Therapy of patients with human T-cell lymphotrophic virus I-induced adult T-cell leukemia with anti-Tac, a monoclonal antibody to the receptor for interleukin-2. Blood. 1988 Nov;72(5):1805-16. PMID 2846094
- [Background] Waldmann TA, White JD, Goldman CK, Top L, Grant A, Bamford R, Roessler E, Horak ID, Zaknoen S, Kasten-Sportes C, et al. The interleukin-2 receptor: a target for monoclonal antibody treatment of human T-cell lymphotrophic virus I-induced adult T-cell leukemia. Blood. 1993 Sep 15;82(6):1701-12. PMID 8400227
- [Background] Gill PS, Harrington W Jr, Kaplan MH, Ribeiro RC, Bennett JM, Liebman HA, Bernstein-Singer M, Espina BM, Cabral L, Allen S, et al. Treatment of adult T-cell leukemia-lymphoma with a combination of interferon alfa and zidovudine. N Engl J Med. 1995 Jun 29;332(26):1744-8. doi: 10.1056/NEJM199506293322603. PMID 7760890
- [Background] Thrush GR, Lark LR, Clinchy BC, Vitetta ES. Immunotoxins: an update. Annu Rev Immunol. 1996;14:49-71. doi: 10.1146/annurev.immunol.14.1.49. PMID 8717507
- [Background] Ghetie V, Ghetie MA, Uhr JW, Vitetta ES. Large scale preparation of immunotoxins constructed with the Fab' fragment of IgG1 murine monoclonal antibodies and chemically deglycosylated ricin A chain. J Immunol Methods. 1988 Sep 13;112(2):267-77. doi: 10.1016/0022-1759(88)90367-5. PMID 3262139
- [Background] Barth S, Schnell R, Diehl V, Engert A. Development of immunotoxins for potential clinical use in Hodgkin's disease. Ann Oncol. 1996;7 Suppl 4:135-41. doi: 10.1093/annonc/7.suppl_4.s135. PMID 8836425
- [Background] Winkler U, Gottstein C, Schon G, Kapp U, Wolf J, Hansmann ML, Bohlen H, Thorpe P, Diehl V, Engert A. Successful treatment of disseminated human Hodgkin's disease in SCID mice with deglycosylated ricin A-chain immunotoxins. Blood. 1994 Jan 15;83(2):466-75. PMID 8286745
- [Background] Engert A, Diehl V, Schnell R, Radszuhn A, Hatwig MT, Drillich S, Schon G, Bohlen H, Tesch H, Hansmann ML, Barth S, Schindler J, Ghetie V, Uhr J, Vitetta E. A phase-I study of an anti-CD25 ricin A-chain immunotoxin (RFT5-SMPT-dgA) in patients with refractory Hodgkin's lymphoma. Blood. 1997 Jan 15;89(2):403-10. PMID 9002941
- [Background] Schnell R, Vitetta E, Schindler J, Borchmann P, Barth S, Ghetie V, Hell K, Drillich S, Diehl V, Engert A. Treatment of refractory Hodgkin's lymphoma patients with an anti-CD25 ricin A-chain immunotoxin. Leukemia. 2000 Jan;14(1):129-35. doi: 10.1038/sj.leu.2401626. PMID 10637488
- [Background] Martin PJ, Pei J, Gooley T, Anasetti C, Appelbaum FR, Deeg J, Hansen JA, Nash RA, Petersdorf EW, Storb R, Ghetie V, Schindler J, Vitetta ES. Evaluation of a CD25-specific immunotoxin for prevention of graft-versus-host disease after unrelated marrow transplantation. Biol Blood Marrow Transplant. 2004 Aug;10(8):552-60. doi: 10.1016/j.bbmt.2004.04.002. PMID 15282533
- [Background] Amrolia PJ, Mucioli-Casadei G, Huls H, Heslop HE, Schindler J, Veys P, Vitetta ES, Brenner MK. Add-back of allodepleted donor T cells to improve immune reconstitution after haplo-identical stem cell transplantation. Cytotherapy. 2005;7(2):116-25. doi: 10.1080/14653240510018181. PMID 16047416

RESULTS

PARTICIPANT FLOW:
Groups:
- Anitbody Therapy: Treatment with Imtox-25 intravenously over 4 hours every other day for 4 doses. Hospital admission is required during this treatment.
  IMTOX-25: This agent is supplied as a sterile solution at 0.5 mg/ml. Thus a vial with 5 mls contains 2.5 mg IMTOX-25 15 mg/m²/cycle IV; The calculated total dose for the cycle will be divided by four and given on Days 1, 3, 5 and 7.
  IMTOX-25: Imtox-25 is an immunotoxin. It is an antibody that is bound to a piece of the poison ricin. This antibody have been shown to bind to leukemia cells and kill them because of the ricin.
Period: Overall Study
Arm/Group | Anitbody Therapy
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Only 1 patient was enrolled prior to study termination.
Arm/Group | Anitbody Therapy
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Response of Imtox-25
Description: To determine any anti-tumor activity of Imtox-25 in relapsed/refractory ATL patients within the confines of a Phase II study as defined by overall response
Time Frame: 28 days
Population: Data was not collected and/or aggregated and therefore not analyzed for the 1 patient on this study.
Arm/Group | Anitbody Therapy
Number analyzed (Participants) | 0

2. Secondary Outcome: Toxicity and Affect of Treatment
Description: To determine the toxicity of Imtox-25 in ATL patients To measure levels of human anti-mouse (HAMA) and human anti-dgA (HARA) antibodies.
  To determine whether the expression of the CD25 cell surface antigens is affected by treatment with Imtox-25 using flow cytometric analysis of lymphoblasts in peripheral blood and bone marrow
Time Frame: 28 days +
Population: Data was not collected and/or aggregated and therefore not analyzed for the 1 patient on this study.
Arm/Group | Anitbody Therapy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 28 days
Arm/Group | Anitbody Therapy
All-Cause Mortality (participants affected / at risk) | 1/1
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anitbody Therapy (N=1)
Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes